CLINICAL TRIAL: NCT04957953
Title: Prospective Cohort of Pregnant Women Vaccinated Against Covid-19.
Brief Title: Pregnant Women Vaccinated Against Covid-19.
Acronym: COVACPREG
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0627; 2021-A01523-38 (Other: ID-RCB)
Record Dates: First submitted 2021-07-07; First posted 2021-07-12 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Pregnant Women Vaccinated Against Covid-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant Women Vaccinated against Covid-19: Woman over 18 years of age who has received at least one Covid-19 vaccine during her pregnancy, regardless of the trimester of pregnancy.
  Interventions: Other: Patient's consent; Other: Inclusion form; Other: Adverse reaction report form.; Diagnostic Test: Follow-up report form.

INTERVENTIONS:
Other: Patient's consent — Primary enrolment will be carried out at the time of vaccination at the main vaccination sites, with the patient's consent. The agreement form filled in online includes the surname, first name, month and year of birth. This form serves as an agreement to participate in the study.
Other: Inclusion form — This form includes the date of the last menstrual period, vaccination data (type of vaccine, date of vaccination, 1st or 2nd injection, etc.), socio-demographic data of the pregnant woman, medical and surgical history, gynaecological and obstetrical history, a description of the current pregnancy, and the medication taken by the patient during her pregnancy....
  A link to complete this form (with the unique identifier) will be sent to each woman included who has given her consent to participate.
Other: Adverse reaction report form. — One month after each injection of the vaccine, information will be collected on any vaccination-related adverse reactions that may impact the pregnancy (fever, hypertension, etc.) or on the onset of a Covid-19 infection,
Diagnostic Test: Follow-up report form. — In the 2 months following the expected delivery date, information will be collected on the outcome of the pregnancy (delivery, spontaneous abortion, etc.) and maternal clinical signs (pre-eclampsia, gestational hypertension, gestational diabetes, etc.). Before sending the link to this form, information will be sent to the second holder of parental authority. In the absence of opposition, data on the newborn will be collected (sex, height, weight, head circumference, Apgar, malformation, neonatal pathology, etc.)

SUMMARY:
Establish a cohort of pregnant women exposed to a COVID19 vaccine, whether or not they have experienced an adverse event, to assess the potential effects of vaccines on the course of pregnancy, on the fetus or newborn and on the mother.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years and over,
* Pregnant,
* Vaccinated against COVID-19,
* Not having expressed any objection to inclusion in the cohort

Exclusion Criteria:

* No agreement at inclusion,
* Age under 18 years

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Any pregnant woman who has received at least one Covid-19 vaccine during her pregnancy, regardless of the trimester of pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 1393 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
To assess the potential effects of vaccines on the course of pregnancy. | One month after injection
  Pregnancy outcomes including the rate of spontaneous miscarriage, fetal death in utero, stillbirth
To assess the potential effects of vaccines on the fetus or newborn | One month after injection
  Characteristics of newborns (weight, height etc.) Malformation rate
To assess the potential effects of vaccines on the mother. | One month after injection
  Rates and types of adverse events following vaccination in pregnant women vaccinated against COVID 19

CONTACTS AND LOCATIONS:
Overall Officials: Judith COTTIN, Principal Investigator — Service Hospitalo-Universitaire de Pharmacotoxicologie
Locations (1):
- Service Hospitalo-Universitaire de Pharmacotoxicologie, Lyon, France